CLINICAL TRIAL: NCT00005548
Title: Green Tea Consumption and Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5092; R03HL062577 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-01

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To examine the prospective association of green tea consumption to the incidence and mortality of coronary heart disease (CHD) using multivariate analysis while controlling for the potential confounding effects of cholesterol, triglycerides, glucose and dietary nutrients.

DETAILED DESCRIPTION:
BACKGROUND:

Both in vivo and in vitro experiments have show that flavonoids, antioxidants which are rich in green tea, are potentially as beneficial as vitamin E, beta-carotene and vitamin C in reducing the risk of cardiovascular disease. Thus, the possible preventive effects of green tea on CHD have begun to raise research interests in green tea sufficiently to inquire about its beneficial effects formally in humans. However, few epidemiologic studies have been carried out to directly examine the effects of green tea on CHD. The Honolulu Heart Program (HHP) is a 30 year longitudinal study of CHD and stroke among 8,006 Japanese American men living on Oahu Hawaii. Until the end of 1992, 1,888 men from this cohort were defined as having incident CHD; this includes 396 deaths due to CHD. The baseline examination for the HHP was conducted during 1965-68. A comprehensive physical examination and 24 hour dietary recall interview were administered. Within the original cohort more than 75 percent men reported to have drunk green tea daily. The amount consumed per day varied considerably from low to high doses. The high prevalence of green tea consumption coupled with dose information (i.e low, moderate and high consumption) provides good opportunities to examine the relationships of green tea consumption and CHD.

DESIGN NARRATIVE:

The study uses the Honolulu Heart Program data to examine the prospective association of green tea consumption to the incidence and mortality of CHD using multivariate analysis while controlling for the potential confounding effects of cholesterol, triglycerides, glucose and dietary nutrients.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-04; Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boji Huang — University of Toledo